CLINICAL TRIAL: NCT05488756
Title: Comparison of Three Different Exercise Training in Patients With Chronic Neck Pain: A Randomized Study
Brief Title: Comparison of the Different Exercises on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Clinical investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neck Pain
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Neck Pain; Pain, Neck
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Conventional training plus isometric neck exercises
  Interventions: Other: Group 1
- Group 2 (Experimental): Conventional training plus deep cervical flexor exercises
  Interventions: Other: Group 2
- Group 3 (Experimental): Conventional training plus stabilization exercises of the neck and core region
  Interventions: Other: Group 3

INTERVENTIONS:
Other: Group 1 — Physical therapy agents and isometric exercise training will be applied to the patients. These will be administered a combination of transcutaneous electrical nerve stimulation, ultrasound, a hot pack, and isometric training 3 times a week for 4 weeks by the physical therapist.
  Arms: Group 1
Other: Group 2 — Physical therapy agents and deep cervical flexor muscle training will be applied to the patients. These will be administered a combination of transcutaneous electrical nerve stimulation, ultrasound, a hot pack, and muscle training 3 times a week for 4 weeks by the physical therapist. Training of the craniocervical flexor muscles is going to be focused on the deep flexor muscles such as longus capitis and longus colli muscles, making neck flexion, not the head.
  Arms: Group 2
Other: Group 3 — Physical therapy agents and core stabilization training will be applied to the patients. These will be administered a combination of transcutaneous electrical nerve stimulation, ultrasound, a hot pack, and stabilization training 3 times a week for 4 weeks by the physical therapist. These exercises will be performed for 10 repetitions with 10 seconds of contraction and 5 seconds of relaxation.
  Arms: Group 3

SUMMARY:
Neck pain is a widespread problem in the general population and is second only to low back pain in musculoskeletal issues.

DETAILED DESCRIPTION:
The aim of this study is to compare the conventional therapy, cervical stabilization exercise approach, and core stabilization exercise in addiction to cervical stabilization in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain more than 3 months
* Medically stable

Exclusion Criteria:

* Patients with benign or tumors in the cervical region
* Patients with active, localized osseous and discal infection in the spine (spondylodiscitis)
* Patients with history of spinal fractures
* Patients with congenital anomaly
* Patients with neck surgery and spinal instability

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Assessment | 4 weeks
  The 11-point Verbal Numeric Pain Scale (VNPS; 0 means no pain; 10 means worst pain) will be use to assess pain intensity. The VNPS is a reliable and valid measure for subjective pain measurement. Participants will be asked to report the pain severity at that moment on a scale from 0 to 10.

SECONDARY OUTCOMES:
Demografic Characteristic of Participants | 1 week before the first treatment session
  The general demographic information of participants such as gender, age, body mass index will be recorded in a form created by investigators. Body mass index (BMI) values will be calculated by dividing body weights by the square of the height and be expressed in kg/m2.
Posture Evaluation | 4 weeks
  Reedco's posture score will be used in posture evaluation. The score is a standard tool and it is administered by visual inspection of 10 postural traits viewed laterally (sagittal view including neck, upper back, trunk, abdomen, and lower back) or from behind (coronal view including head, shoulders, spine, hips, and ankles). The scores are marked as follows: a value of 0 equals poor posture or severe deviation, a value of 5 equals fair posture or minimal to moderate deviation, and a value of 10 equals good posture or normal alignment. The maximum score of 100 indicates good posture and a score of 59% or less is recorded as postural dysfunction.
Evaluation of Cervical Range of Motion | 4 weeks
  Cervical ROM will be evaluated using a goniometer while the patient sitting on the chair with both feet on the ground. In the evaluation, after the goniometer is brought to the neutral position, the patient is asked to perform the desired movement with the head: flexion, extension, right and left lateral flexion, right and left rotation. A degree will be recorded for each neck motion and be used in the average analysis
Disability Evaluation | 4 weeks
  Neck Disability Index will be used to evaluate daily activities and ability. The form contains of 10 questions related to pain intensity, lifting, concentration, reading, headache, self-management, driving, working, sleeping, and daily activities. The score of each question is 0-5 according to the options and the total score is recorded by adding the scores of all answers. The lower the total score of the test, the less the effect of pain on performance in daily activities. The higher the score, the greater the performance of daily activities is affected.
Assessment of Quality of Life | 4 weeks
  The Short Form-36 is a test that includes a 36-item self-administered comprehensive health status questionnaire and will be used to assess the quality of life. This test includes questions evaluating physical function, social function, limitations due to physical health, limitations due to mental health, vitality, body pain, and general health. In this test, two scores are generally calculated, the combined physical and mental summary score. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Eylül Pınar Kısa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No